CLINICAL TRIAL: NCT00675259
Title: Phase II Trial of Neoadjuvant Chemotherapy [NCT] With Weekly Nanoparticle Albumin-bound Paclitaxel [Nab-paclitaxel; Abraxane®] in Combination With Carboplatin and Bevacizumab in Women With Clinical Stages I-III Breast Cancer
Brief Title: Phase II NCT (Neoadjuvant Chemotherapy) w/ Weekly Abraxane in Combination With Carboplatin & Bevacizumab in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-07074; NCI-2011-03188 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2008-05-08; First posted 2008-05-09 (Estimated); Results first posted 2016-08-24 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Surgical Procedures, Operative; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant, Surgery, Adjuvant (Experimental): Neoadjuvant chemotherapy : Nab-paclitaxel and carboplatin on days 1, 8, and 15 in combination with bevacizumab on days 1 and 15 administered every 28 days for 5 cycles followed by 1 cycle with Nab-paclitaxel and carboplatin on days 1, 8, and 15. Definitive surgery with either lumpectomy or mastectomy along with axillary lymph node dissection for all pre neo adjuvant chemotherapy node-positive patients approximately 4-5 weeks after the completion of NCT. Use of additional adjuvant chemotherapy and/or radiation therapy depends upon the treating physicians' judgment. Radiation therapy should begin no sooner than 6 weeks after breast cancer surgery. All hormone receptor positive patients will receive endocrine therapy. All patients will receive 6 months of adjuvant bevacizumab every 3 weeks. If using an adjuvant anthracycline-containing regimen then bevacizumab will be administered ≥ 3 weeks after completing the regimen.
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: nab-paclitaxel; Procedure: Surgery; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: bevacizumab — bevacizumab 10 mg/kg on days 1 and 15 administered every 28 days [1 cycle] for 5 cycles
  Other Names: Avastin
Drug: carboplatin — AUC 2 IV on days 1, 8, and 15
  Other Names: Paraplatin; Paraplatin-AQ
Drug: nab-paclitaxel — 100 mg/M2 IV
  Other Names: Abraxane
Procedure: Surgery — lumpectomy or mastectomy along with axillary lymph node dissection approximately 4-5 weeks after completion of NCT.
Drug: Adjuvant chemotherapy — All hormone receptor positive patients will receive endocrine therapy. All patients will receive 6 months of adjuvant bevacizumab at 15 mg/kg IV every 3 weeks. If using an adjuvant anthracycline-containing regimen then bevacizumab will be administered ≥ 3 weeks after completing the regimen.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel albumin-stabilized nanoparticle formulation and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some find tumor cells and help kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Bevacizumab may also stop the growth of breast cancer by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving bevacizumab after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying the side effects and how well giving paclitaxel albumin-stabilized nanoparticle formulation and carboplatin together with bevacizumab works in treating women undergoing surgery for stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete pathological response (pCR) in the breast/axillary lymph nodes in women with stage II or III breast cancer treated with neoadjuvant therapy comprising paclitaxel albumin-stabilized nanoparticle formulation, carboplatin, and bevacizumab followed by surgery and adjuvant bevacizumab.
* To determine the side effects of this regimen in these patients.

Secondary

* To evaluate dynamic contrast-enhanced magnetic resonance imaging in assessing pCR.
* To measure LZTS1 gene expression before and after neoadjuvant therapy to evaluate whether LZTS1 gene expression correlates with pCR.
* To evaluate the feasibility and toxicity of adjuvant bevacizumab when administered for 6 months.

OUTLINE:

* Neoadjuvant therapy: Patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 30 minutes on days 1, 8, and 15 and bevacizumab IV over 30-90 minutes on days 1 and 15. Treatment repeats every 28 days for 5 courses. After completion of course 5, patients receive paclitaxel albumin-stabilized nanoparticle formulation IV over 30 minutes and carboplatin IV over 30 minutes on days 1, 8, and 15. Patients then proceed to surgery.
* Surgery: Approximately 4-5 weeks after completion of neoadjuvant therapy, patients undergo definitive surgery (either lumpectomy or mastectomy). Patients with node-positive disease or inflammatory breast cancer at baseline also undergo axillary lymph node dissection. Patients then proceed to adjuvant therapy.
* Adjuvant therapy: Beginning approximately 6 weeks after surgery, patients receive bevacizumab IV over 30-90 minutes once every 3 weeks for 6 months. Patients with hormone receptor-positive disease also receive endocrine therapy. Patients may also receive additional adjuvant chemotherapy or radiotherapy at the discretion of the treating physician.

Patients undergo dynamic contrast-enhanced magnetic resonance imaging at baseline, after course 2 of neoadjuvant therapy, and after completion of neoadjuvant therapy (prior to definitive surgery) for assessment of tumor response. Tumor tissue is collected at baseline and during surgery for correlative laboratory studies. LZST1 gene expression is assessed by immunohistochemistry before and after neoadjuvant therapy.

ELIGIBILITY:
Inclusion:

* Histologically confirmed breast cancer
* Clinically or radiographically measurable residual tumor after core biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Age ≥18 yrs
* Absolute neutrophil count ≥ 1,500/mm³
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100,000/ mm³
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Urine protein:creatinine ratio < 1.0
* AST (aspartate aminotransferase) and ALT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin normal
* Women of childbearing potential must use effective contraception
* Left ventricular ejection fraction (LVEF) normal by echocardiogram or MUGA

Exclusion:

* No residual tumor after initial biopsy
* Peripheral neuropathy of grade 2 or higher
* HER-2 neu overexpression either by IHC 3+ or FISH+
* No history of any prior treatment of breast cancer.
* No history of unstable angina or myocardial infarction within the past 12 months
* Pregnant or nursing women
* Anticoagulation therapy within the last 6 months
* History of gastrointestinal bleeding
* Recent hemoptysis
* No known hepatitis B or HIV seropositivity
* No inadequately controlled hypertension, defined as systolic blood pressure (BP) > 150 mm Hg and/or diastolic BP > 100 mm Hg despite antihypertensive medications
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association class II-IV congestive heart failure
* History of stroke or transient ischemic attack at any time
* Significant vascular disease (e.g., aortic aneurysm or aortic dissection)
* No symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Significant traumatic injury within the past 28 days
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* Serious, non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Mrozek, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Mrozek E, Layman R, Ramaswamy B, Lustberg M, Vecchione A, Knopp MV, Shapiro CL. Phase II trial of neoadjuvant weekly nanoparticle albumin-bound paclitaxel, carboplatin, and biweekly bevacizumab therapy in women with clinical stage II or III HER2-negative breast cancer. Clin Breast Cancer. 2014 Aug;14(4):228-34. doi: 10.1016/j.clbc.2014.02.005. Epub 2014 Feb 20. PMID 24703985
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant, Surgery, Adjuvant: Neoadjuvant chemotherapy : Nab-paclitaxel and carboplatin on days 1, 8, and 15 in combination with bevacizumab on days 1 and 15 administered every 28 days for 5 cycles followed by 1 cycle with Nab-paclitaxel and carboplatin on days 1, 8, and 15. Definitive surgery with either lumpectomy or mastectomy along with axillary lymph node dissection for all pre neo adjuvant chemotherapy node-positive patients approximately 4-5 weeks after the completion of NCT (Neoadjuvant chemotherapy). Use of additional adjuvant chemotherapy and/or radiation therapy depends upon the treating physicians' judgment. Radiation therapy should begin no sooner than 6 weeks after breast cancer surgery. All hormone receptor positive patients will receive endocrine therapy. All patients will receive 6 months of adjuvant bevacizumab every 3 weeks. If using an adjuvant anthracycline-containing regimen then bevacizumab will be administered ≥ 3 weeks after completing the regimen.
Period: Overall Study
Arm/Group | Neoadjuvant, Surgery, Adjuvant
Started | 33
Completed | 19
Not Completed | 14

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant, Surgery, Adjuvant
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 48 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 33
Menopausal status [Number; unit: patients]
  Premenopausal | 21
  Postmenopausal | 12
Receptor status (all HER2/neu negative) [Number; unit: patients] — ER=estrogen receptor HER2/neu=human epidermal growth factor receptor 2 PR=progesterone receptor
  patients
    Triple negative | 12
    ER and PR positive | 21
Axillary lymph node status before NCT [Number; unit: patients] — NCT=neoadjuvant chemotherapy SLNB=sentinel lymph node biopsy
  patients
    Positive by core biopsy | 15
    Positive by SLNB | 4
    Negative by core biopsy | 5
    Negative by SLNB | 8
    Not evaluated | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pathologic Complete Response (pCR)
Description: pCR was defined as the absence of viable invasive tumor cells in the surgical breast specimen and axillary lymph nodes.
Time Frame: every 4 weeks
Population: Includes patients with triple negative breast cancer and ER+/PR+ breast cancer.
Measure: Number; unit: patients
Arm/Group | Neoadjuvant, Surgery, Adjuvant
Number analyzed (Participants) | 33
patients | 6

2. Primary Outcome: Side Effects of Weekly Nab-paclitaxel, Carboplatin and Bevacizumab
Description: Adverse events were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 3.0
Time Frame: Up to 4 weeks
Population: all grade 3 adverse events
Measure: Number; unit: patients
Groups:
- Adjuvant Bevacizumab: Patients received 6 months of adjuvant bevacizumab therapy
Arm/Group | Adjuvant Bevacizumab
Number analyzed (Participants) | 33
patients
  hypersensitivity reaction | 1
  hypertension | 2
  infection at mastectomy site | 1

3. Secondary Outcome: Evaluation of Dynamic Contrast-enhanced Magnetic Resonance Imaging in Assessing pCR at Baseline and After 2 Cycles of Neoadjuvant Therapy
Description: Relative angiogenic volume (AV) was defined as the ratio of AV to the geometric volume of the tumor in the breast.
Time Frame: after 2 cycles of therapy
Population: Data only available for 20 of the 28 evaluable patients
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Neoadjuvant, Surgery, Adjuvant
Number analyzed (Participants) | 20
ratio
  Baseline DCE-MRI | 0.65 (0.18)
  Relative AV at end of cycle 2 | .4 (.33)

4. Secondary Outcome: Overall Expression of LZTS1 Before and After Neoadjuvant Therapy as Assessed by Immunohistochemistry
Description: LZTS1 expression in breast cancer cells collected prior to NCT
Time Frame: prior to surgery
Population: LZTS1 expression in breast cancer cells collected prior to NCT was assessed in 27 patients who had evaluable core biopsies.
Measure: Number; unit: patients
Groups:
- Patients With TNBC: Women with triple negative breast cancer (TNBC)
- Patients With pCR: Pathologic complete response (pCR)
- Patients With Hormone-responsive BC: Hormone-responsive breast cancer (BC)
Arm/Group | Patients With TNBC | Patients With pCR | Patients With Hormone-responsive BC
Number analyzed (Participants) | 11 | 5 | 16
patients
  0 | 2 | 2 | 6
  +1 | 0 | 0 | 2
  +2 | 3 | 2 | 2
  +3 | 6 | 1 | 6

ADVERSE EVENTS:
Description: The NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 was used for grading patients adverse events.
Arm/Group | Toxicities During Neoadjuvant Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 33/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Toxicities During Neoadjuvant Chemotherapy (N=33)
Leukopenia (Blood and lymphatic system disorders) | 26 (26)
Anemia (Blood and lymphatic system disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 29 (29)
Wound Complications (Injury, poisoning and procedural complications) | 3 (3)
Fatigue (General disorders) | 28 (28)
Nausea (Gastrointestinal disorders) | 8 (8)
Infection with normal ANC (Infections and infestations) | 8 (8)
Peripherial neuropathy (Nervous system disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 8 (8)
Hypertension (Vascular disorders) | 6 (6)
Depressed Mood (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 12 (12)
Headache (Nervous system disorders) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Mucositis (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes